CLINICAL TRIAL: NCT04705207
Title: Exploratory Study of the Impact of Foot Reflexology on Chronic Pain in Parkinsonian Patients
Brief Title: Foot Reflexology on Chronic Pain in Parkinsonian Patients
Acronym: DOREPAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RC 31/20/0279
Record Dates: First submitted 2021-01-05; First posted 2021-01-12 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease
Keywords: Pain; Foot Reflexology
MeSH Terms: conditions — Parkinson Disease; Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: a group has intervention, a group has placebo intervention
Who Masked: Participant, Outcomes Assessor
Masking Description: placebo is a traditional massage instead of a intervention reflexology massage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reflexology massage (Experimental): foot reflexology massage
  Interventions: Procedure: reflexology massage
- sham massage (Placebo Comparator): traditional foot massage
  Interventions: Procedure: sham massage

INTERVENTIONS:
Procedure: reflexology massage — the patient receive only foot reflexology massage
  Arms: reflexology massage
Procedure: sham massage — the patient receive only foot traditional massage
  Arms: sham massage

SUMMARY:
Pain is one of the non-motor symptoms of Parkinson's disease still poorly known and misdiagnosed and its management is complex. This encourage to explore new non-drug therapeutic paths, such as foot reflexology (FR). the present study proposed a comparison of the evolution of different parameters, quantitative and qualitative, to identify biomarkers and highlight the specific effect of FR on pain, compared to sham massage.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disease characterized by the destruction of specific neurons population involved in movement control. Pain is one of the non-motor symptoms still poorly known and misdiagnosed. In addition to this fact, its management is complex. At present, the medical community has no effective solution to reduce pain to an acceptable level in terms of intensity or frequency.

Pain is a personal, subjective experience with an affective and cognitive dimension. The context and its psychological impact can amplify as well as alleviate the pain. Thus, non-pharmacological treatment (NPT) that influence the psychological state (mood, level of stress, ...) can also modulate the pain experience through the brain matrix of pain. Among them, foot reflexology, which by stimulating reflex zones located on the feet, makes it possible to modify the perception of the pain and to modify the subjective / emotional valence of the pain. In this study, we propose to evaluate this technique, by postulating that it should reduce the chronic pain of patients with Parkinson's disease.

This project is innovative and original in two dimensions : On the one hand, the pain of patients in PD is still often underestimated, there is in the mere fact of devoting a study a real dynamic of change in the consideration of the patients concerned and in the management of this non-motor symptom. On the other hand, the increasing use of NPT requires that clinical studies be conducted. To date, it is clear that very few or no reliable studies have been conducted on the subject. We wish to develop complementary non-pharmacological management to provide concrete help to Parkinson's patients and thus initiate the scientific validation of NPT as recommended by the High Authority of Health.

The study hypothesize that through a comparison of the evolution of different parameters, quantitative and qualitative, this study will allow to identify biomarkers and highlight the specific effect of FR on pain, compared to sham massage.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an age egal at 18 years old or more,
* Patient presenting a little fluctuating Parkinson's disease attested by a score ≤ 2 on the MDS UPDRS IV,
* Patients with chronic pain for at least 3 months with a VAS ≥ 4
* Patients whose anti-parkinsonian treatment is stable throughout the duration of the study and at least for 4 weeks.

Exclusion Criteria:

* Patients with cognitive impairment defined by an MOCA<25
* Patient presenting contraindication to carrying out the MRI examination
* Patient refusing to be informed of any abnormality detected on brain MRI
* Patient included in a clinical trial that potentially interferes with the objective of the study,
* Patient resistant to foot massage,
* Patient having benefited from a Foot reflexology session in the last 6 months, - Patient presenting skin lesions in the feet,
* Patient having a recent fracture in the feet,
* Patient having an history of phlebitis less than 3 months and history of deep vein thrombosis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
evaluation of changes in the mean intensity of chronic pain | Day 1 and week 12
  Visual Analog Scale (VAS) ok pain (0 is no pain, 10 is the most high pain)

SECONDARY OUTCOMES:
evaluation of the change in pain on the VAS | Day 1, week 3, week 6, week 9 and week 12
  Visual Analog Scale of change of pain (0 is no pain, 10 is the most high pain)
evaluation of change in chronic pain | Day 1 and week 12
  King's Parkinson's disease Pain Scale (KPPS)
evaluation of change in chronic pain | Day 1 and week 12
  Brief Pain Inventory (BPI)
evaluation of change in chronic pain | Day 1 and week 12
  Primary Parkinsonian Pain Diagnostic Questionnaire (3PDQ)
evaluation of the consumption of analgesics | Day 1, week 3, week 6, week 9 and week 12
  completion by the patient of a logbook of analgesic treatments
evaluation of anxiety and depression | Day 1 and week 12
  Hospital Anxiety Depression (HAD) scale
connectivity of brain networks | Day 1 and week 12
  observation of connectivity cards by Functional Magnetic Resonance Imaging (MRI)
evaluation of the threshold of perception of subjective warm pain | Day 1, week 9 and week 12
  contact thermode is used to dermine the threshold of perception

CONTACTS AND LOCATIONS:
Overall Officials: Christine BREFEL-COURBON, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

REFERENCES:
- [Derived] Boussac M, Harroch E, Joineau K, Descamps E, Brefel-Courbon C. Neuro-functional correlates of personality dimensions in Parkinson's disease. Front Pharmacol. 2025 Nov 7;16:1705937. doi: 10.3389/fphar.2025.1705937. eCollection 2025. PMID 41282613
- [Derived] Joineau K, Harroch E, Boussac M, Fabbri M, Leung C, Ory-Magne F, Rousseau V, Peran P, Brefel-Courbon C, Descamps E. Effect of foot reflexology on chronic pain in Parkinson's disease: A randomized controlled trial. PLoS One. 2025 Jul 28;20(7):e0327865. doi: 10.1371/journal.pone.0327865. eCollection 2025. PMID 40720491